CLINICAL TRIAL: NCT06692608
Title: Effects of an Isometric Training Session on Post-exercise Neuromuscular Function When Compared to a Dynamic Strength Training Session in Youth Soccer Players
Brief Title: Effects of an Isometric Training Session on Post-exercise Neuromuscular Function When Compared to Dynamic Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ST_002
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Strength Training Effects
Keywords: strength; isometric; dynamic; soccer
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic strength training (Active Comparator)
  Interventions: Other: strength training
- Isometric strength training (Experimental)
  Interventions: Other: strength training

INTERVENTIONS:
Other: strength training — Comparison between isometric and dynamic strength training in soccer players

SUMMARY:
The existing literature shows that maximum strength can be improved through both dynamic and isometric strength training. However, there is a perception that dynamic training has a negative effect on short-term neuromuscular performance in soccer players. Hence, the aim of this study was to compare the neuromuscular impairment after isometric and dynamic training sessions in young soccer players.

ELIGIBILITY:
Inclusion Criteria:

* soccer players
* Competing at national level

Exclusion Criteria:

* Injured or recently injured athletes

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
countermovement jump | baseline (pre-test), 30 minutes and 24 hours post intervention
bar velocity | baseline (pre-test), 30 minutes and 24 hours post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided